CLINICAL TRIAL: NCT04859946
Title: Itacitinib to Prevent Graft Versus Host Disease
Brief Title: Itacitinib for the Prevention of Graft Versus Host Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0971; NCI-2021-02784 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0971 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Hematologic and Lymphocytic Disorder
MeSH Terms: conditions — Hematologic Diseases | interventions — Stem Cell Transplantation; Busulfan; Cyclophosphamide; fludarabine; itacitinib; INCB039110; Tacrolimus; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (itacitinib) (Experimental): CONDITIONING: Patients receive busulfan IV over 3 hours on days -20, -13, and -6 to -3, thiotepa IV on day -7, and fludarabine IV over 1 hour on days -6 to -3.
  STEM CELL TRANSPLANT: Patients undergo stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days 3 and 4. Patients also receive itacitinib PO QD on days 5-60 in the absence of disease progression or unacceptable toxicity. Beginning day 5 after stem cell transplant, patients also receive tacrolimus IV over 24 hours until able to tolerate oral tacrolimus, whereby patients then receive tacrolimus PO BID.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Itacitinib; Drug: Tacrolimus; Drug: Thiotepa

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo stem cell transplant
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Itacitinib — Given PO
  Other Names: INCB 039110; INCB-039110; INCB039110
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Thiotepa — Given IV
  Other Names: 1,1'',1''''-Phosphinothioylidynetrisaziridine; Girostan; N,N'', N''''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312

SUMMARY:
This phase II trial studies if itacitinib plus standard of care treatment may help prevent graft-versus-host-disease (GVHD) in patients who have received an allogeneic (donor) stem cell transplant. An allogeneic transplant uses blood-making cells from a family member or unrelated donor to remove and replace a patient's abnormal blood cells. Sometimes the transplanted cells from a donor can attack the body's normal cells (called graft-versus-host disease). Giving itacitinib with standard of care treatment after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the 100-day acute grade 2-4 GvHD rate to matched controls.

SECONDARY OBJECTIVES:

I. To compare the 1-year rate of GvHD-free, relapse-free survival to matched controls.

II. To assess the time to neutrophil and platelet engraftment. III. To assess the toxicity profile associated with this regimen. IV. To assess the incidence of severe grade 3-4 acute GVHD. V. To assess the incidence of limited, extensive, and moderate to severe chronic GVHD.

VI. To assess the incidence of disease relapse. VII. To assess the incidence of non-relapse mortality. VIII. To assess overall survival and progression-free survival. IX. To assess immunosuppression discontinuation rate.

TERTIARY OBJECTIVE (CORRELATIVE STUDY):

I. Immune recovery and cytokines at various time points pre- and post- transplant

OUTLINE:

CONDITIONING: Patients receive busulfan intravenously (IV) over 3 hours on days -20, -13, and -6 to -3, thiotepa IV on day -7, and fludarabine IV over 1 hour on days -6 to -3.

STEM CELL TRANSPLANT: Patients undergo stem cell transplant on day 0.

GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days 3 and 4. Patients also receive itacitinib orally (PO) once daily (QD) on days 5-60 in the absence of disease progression or unacceptable toxicity. Beginning day 5 after stem cell transplant, patients also receive tacrolimus IV over 24 hours until able to tolerate oral tacrolimus, whereby patients then receive tacrolimus PO twice daily (BID).

After completion of study intervention, patients are followed up at days 100, 180, and 365 after stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years to less than or equal to 70 years
* English and non-English speaking patients are eligible
* Karnofsky performance status of at least 70
* Patients with hematological disorders undergoing allogeneic stem cell transplant (ASCT) with conditioning regimen of fractionated busulfan, thiotepa and fludarabine
* Donor will be matched at HLA A, B, C and DR at allele level. Donor will be either HLA-identical sibling or at least 7/8 matched unrelated donor, or a haploidentical related donor available.
* Life expectancy of at least 12 weeks (3 months)
* Direct bilirubin not greater than 1 mg/dL
* Alanine transaminase (ALT) less than or equal 3 x upper limit of normal range
* Creatinine clearance >/= 60 ml/ min
* Diffusing capacity for carbon monoxide (DLCO) 50% of predicted corrected for hemoglobin
* Left ventricular ejection fraction (LVEF) of at least 50%
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form (ICF) until at least 30 days after the last dose of study drug. Recommended methods of birth control are:

  * Hormonal contraception (birth control pills, patches, or rings)
  * Intrauterine device (IUD)
  * Birth control injections
  * Double barrier methods (diaphragm with spermicidal gel or condoms with birth control foam)
  * Sterilization of patient or partner ("tubes tied" or vasectomy)
* Patients enrolled on this study may be enrolled on other IND studies at the discretion of the PI

Exclusion Criteria:

* Patients with acute leukemia in the first complete remission and chronic myeloid leukemia in the first chronic phase during the initial enrollment of 6 patients
* Patients with toxicities (Grade > 1) unresolved from prior treatment (including chemotherapy, targeted therapy, immunotherapy, experimental agents, radiation, or surgery)
* Haploidentical recipients should not have donor-specific antibodies (DSA)
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) > class II
  * Active coronary artery disease
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before transplant, or myocardial infarction within 6 months before transplant
* Patients with active hepatitis B and C
* Patients with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with safety or with obtaining informed consent or compliance with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute grade 2-4 graft versus host disease (GVHD) | At 100 days after stem cell transplant
  The 100-day acute grade 2-4 GvHD rate will be compared between groups using Fisher's exact test. Matched logistic regression techniques will also be considered for this endpoint. The proportion of patients with acute grade 2-4 GVHD at 100 days will be reported, along with the corresponding 95% confidence interval.

SECONDARY OUTCOMES:
GVHD-free relapse-free survival | From day of stem cell transplant to time of grade 3 or 4 acute GVHD or chronic GVHD needing systemic immunosuppression or relapse or death whichever occurs first, assessed at 1 year after stem cell transplant
  Will be compared between groups using the log-rank test. The method of Kaplan and Meier will be used to estimate the distribution of GVHD-free, relapse-free survival. The estimated probability will be reported at 1 year along with a corresponding 95% confidence interval. In addition, Cox proportional hazards regression models will be fit to this endpoint, considering clinical, demographic, and treatment covariates of interest.
Time to neutrophil and platelet engraftment | Up to 365 days after stem cell transplant
  Engraftment is defined as the presence of neutrophil recovery by day 28 post stem cell infusion. Neutrophil recovery is defined as a sustained absolute neutrophil count (ANC) > 0.5 x 10^9/L for three consecutive days.
  Initial platelet recovery is defined as the first date of three consecutive laboratory values obtained for platelet count was >= 20 x 10^9/L AND no platelet transfusions were administered for seven consecutive days immediately preceding this date. Will be calculated from the time of transplant and estimated by the Kaplan-Meier method. Distributions will be compared between patients with matched and mismatched donors via the log-rank test.
Overall survival | From day of stem cell transplant to day of death, assessed up to 365 days after stem cell transplant
  Will be calculated from the time of transplant by the method of Kaplan and Meier. Cox proportional hazards regression analysis will be used to assess the association between these survival parameters and clinical and treatment covariates of interest.
Progression-free survival | From day of transplant to day of death or disease progression, assessed up to 365 days after stem cell transplant
  Will be calculated from the time of transplant by the method of Kaplan and Meier. Cox proportional hazards regression analysis will be used to assess the association between these survival parameters and clinical and treatment covariates of interest.
Time to relapse | Up to 365 days after stem cell transplant
Non-relapse mortality | Up to 365 days after stem cell transplant
  Defined as death from any cause other than relapse disease.
Cumulative incidence of limited, extensive, and moderate to severe chronic GVHD | Up to 365 days after stem cell transplant
  The cumulative incidence of acute and chronic GVHD with the competing risk of relapse and death without relapse will be estimated using the method of Gooley, and the method of Fine and Gray will be used to model the incidence by disease and clinical characteristics of interest.
Incidence of adverse events | Up to 365 days after stem cell transplant
  Descriptive statistics will be used to summarize adverse events. Frequency counts and percentages will also be presented of subjects with serious adverse events and adverse events leading to withdrawal. All other safety parameters will be summarized using descriptive statistics or frequency counts. Graphical summaries will be used where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Uday R Popat, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States